CLINICAL TRIAL: NCT00000716
Title: A Multicenter Trial To Evaluate Oral Retrovir in the Treatment of Children With Symptomatic HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 043; NCI-T88-0191N; Protocol 26,341--08; Project P53; FDA 9C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1990-05

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Administration, Oral; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and tolerance of oral zidovudine (AZT) when given over a period of 24 weeks to children between 3 months and 12 years of age. The effectiveness of AZT in treating HIV infection in infants and children will also be evaluated.

HIV infection in children is most often associated with symptomatic disease and poor prognosis. Treatment with antiviral therapy may be effective in altering the course of the disease and decreasing mortality in these children. AZT has been shown to be effective in certain adult patients with symptomatic HIV infection. It is therefore likely that infected children may also benefit from this treatment.

DETAILED DESCRIPTION:
HIV infection in children is most often associated with symptomatic disease and poor prognosis. Treatment with antiviral therapy may be effective in altering the course of the disease and decreasing mortality in these children. AZT has been shown to be effective in certain adult patients with symptomatic HIV infection. It is therefore likely that infected children may also benefit from this treatment.

The participants receive AZT mixed with juice at a dose dependent on body size every 6 hours for 24 weeks. The children are evaluated weekly for the first 4 weeks, every two weeks for the subsequent 8 weeks, and monthly thereafter. Blood samples are collected periodically and cerebrospinal fluid (CSF) by lumbar puncture on 2 occasions.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Amphotericin B and antituberculosis chemotherapy.
* Children who have advanced lymphocytic interstitial pneumonitis (LIP) who are steroid dependent may remain on such therapy.
* Secondary prophylaxis for Pneumocystis carinii pneumonia (PCP) with careful monitoring for possible toxicity due to combination therapy with zidovudine (AZT).

Concurrent Treatment:

Allowed:

* Blood transfusions for hematologic toxicity.
* Immunoglobulin therapy for development of = or > 3 serious bacterial infections while receiving zidovudine. A serious bacterial infection includes septicemia (not catheter related), pneumonia, meningitis, bone or joint infection, or abscess of the body cavity or internal organ.
* The pathogen must be one of the following organisms:
* Staphylococcus aureus, Streptococcus pyogenes, Escherichia coli, Streptococcus group B, Pseudomonas aeruginosa, Hemophilus influenzae B, and Pneumococcus. Laboratory documentation of the pathogen is required.

Patients must comply with the following:

* Life expectancy of more than 6 months.
* Children must have laboratory evidence of HIV infections as demonstrated by either a positive viral culture or detectable serum p24 antigen or repeated positive test for HIV antibody determined by a federally licensed ELISA test and confirmed by Western blot.
* Children under 15 months of age, who are thought to have acquired HIV through perinatal transmission and whose only laboratory evidence of HIV infection is a positive antibody test, must also have increased immunoglobulin levels and decreased absolute number of CD4+ cells or a decreased helper/suppressor ratio.
* AIDS:
* Must have clinical evidence of HIV infection as demonstrated by the presence of one or more of the indicator diseases as defined in the CDC Surveillance definition for AIDS. (NOTE:
* Children with lymphocytic interstitial pneumonitis are excluded unless they meet at least one of the following conditions:
* an additional AIDS-defining opportunistic infection, recurrent serious bacterial infection, HIV encephalopathy, wasting syndrome, or meet the definition of AIDS related complex (ARC).
* ARC:
* Children who present with at least one of the first three clinical findings and one of any other listed below within 2 months of entry or who present with two of the first three symptoms listed:
* <= 500 CD4 cells/mm3 within 4 weeks of entry, persistent (>= 2 months) or recurrent oral candidiasis despite therapy, diarrhea (defined as >= 3 loose stools per day) that is either persistent or recurrent, hepatomegaly, splenomegaly, cardiomyopathy, nephropathy manifested by nephrotic syndrome without evidence of renal failure, 2 or more episodes of herpes stomatitis within a 1-year period, or 2 or more episodes of recurrent herpes zoster or chronic zoster (defined as = or > 30 days duration regardless of therapy).
* Written informed consent from a parent or guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following will be excluded:

* Any active or chronic opportunistic infection at time of entry requiring acute therapy with experimental agents or agents which may affect zidovudine (AZT) toxicity or safety, nor serious bacterial, fungal, or parasitic infections requiring parenteral therapy at the time of entry.

Concurrent Medication:

Concomitant medications should be kept to a minimum.

Excluded:

* Chronic use of drugs that are metabolized by hepatic glucuronidation, such as acetaminophen.
* Acute therapy for active or chronic opportunistic infection with experimental agents or agents which may affect zidovudine (AZT) toxicity.
* Parenteral therapy for serious bacterial, fungal, or parasitic infections.
* Prophylaxis for Pneumocystis carinii pneumonia (PCP) for children who have not had a previous episode of PCP, oral candidiasis, or otitis media.
* Immunoglobulin therapy. Note: Immunoglobulin therapy may be administered to children who develop = > 3 serious bacterial infections while receiving AZT.

Children with lymphocytic interstitial pneumonitis (LIP) as their only clinical sign of HIV infection will be excluded from the study. Children with any of the following laboratory findings within 2 weeks of entry will be excluded:

* A total bilirubin > 3 times Upper Limit of Normal (ULN).
* SGOT > 5 x Upper Limit of Normal in the presence of an age-adjusted abnormal bilirubin.
* Creatinine clearance < 50 ml/min/1.73 m2.
* White blood cells < 2000 cells/mm3.
* Neutrophils < 800 cells/mm3.
* Hematocrit < 24 percent.
* Hemoglobin < 8.0 g /dl.
* Children who will be unable to be followed by their original study center for the 24 weeks of the study will be excluded.

Prior Medication:

Excluded within 2 weeks of study entry:

* Any other experimental therapy or drugs which cause prolonged neutropenia or significant nephrotoxicity.
* Excluded within 4 weeks of study entry:
* Immunomodulating agents including steroids, interferon, isoprinosine, and interleukin-2.
* Excluded within 2 months of study entry:
* Other antiretroviral agents.
* Note: Children with advanced lymphocytic interstitial pneumonitis (LIP) who are steroid dependent may remain on such therapy.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Immunoglobulin.
* Lymphocyte transfusions for immune reconstitution.
* Excluded within 3 months of study entry:
* Bone marrow transplant.

Active alcohol or drug abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70
Dates: Primary Completion 1991-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfert C, Study Chair
Locations (9):
- United States (9):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] McKinney RE Jr, Wilfert C. Growth as a prognostic indicator in children with human immunodeficiency virus infection treated with zidovudine. AIDS Clinical Trials Group Protocol 043 Study Group. J Pediatr. 1994 Nov;125(5 Pt 1):728-33. doi: 10.1016/s0022-3476(94)70065-6. PMID 7965424
- [Background] McKinney RE Jr, Maha MA, Connor EM, Feinberg J, Scott GB, Wulfsohn M, McIntosh K, Borkowsky W, Modlin JF, Weintrub P, et al. A multicenter trial of oral zidovudine in children with advanced human immunodeficiency virus disease. The Protocol 043 Study Group. N Engl J Med. 1991 Apr 11;324(15):1018-25. doi: 10.1056/NEJM199104113241503. PMID 1672443
- [Background] Connor E. Lymphocyte subset changes in children with advanced symptomatic HIV infection treated with oral zidovudine. Int Conf AIDS. 1990 Jun 20-23;6(2):95 (abstract no FB21)
- [Background] Kavanaugh-McHugh A, Ruff A, Rowe S, Holt E, Modlin J, Maha M, Wilfert C. Cardiac abnormalities in pediatric HIV infection. Int Conf AIDS. 1990 Jun 20-23;6(2):198 (abstract no FB483)
- [Background] McKinney RE, Wilfert CM. The efficacy of oral, intermittent zidovudine (ZDV) in a phase II pediatric trial (AIDS clinical trials group study 043). Int Conf AIDS. 1990 Jun 20-23;6(2):94 (abstract no FB18)
- [Background] McKinney RS. Markers prognostic for survival in zidovudine treated, HIV infected children. ACTG Protocol 043 Study Group. American Pediatric Society 104th annual meeting and Society for Pediatric Research 63rd annual meeting; 1994 May 2-5; Seattle. Pediatr AIDS HIV Infect. 1994 Oct;5(5):323 (unnumbered abstract)